CLINICAL TRIAL: NCT04193124
Title: Clinical Implication of Prolonged Vasospasm in Subarachnoid Hemorrhage
Brief Title: Prolonged Vasospasm in Subarachnoid Hemorrhage
Acronym: PVE
Status: Completed | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit at Hospital El Cruce, Hospital El Cruce
Other Study IDs: HEC
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Subarachnoid Hemorrhage; Vasospasm, Intracranial
Keywords: Subarachnoid Hemorrhage; Vasospasm, Intracranial; Transcranial doppler
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prolonged vasospasm: Adult patients with a diagnosis of subarcnoid hemorrhage CT scan or presence of blood in the cerebrospinal fluid were incorporated. Patients with vasospasm were followed daily with transcranial doppler. Prolonged vasospasm was defined for patients who persisted with vasospasm after day 21 of cerebral bleeding.
  Interventions: Diagnostic Test: transcranial doppler.

INTERVENTIONS:
Diagnostic Test: transcranial doppler. — Daily monitoring of transcranial doppler until the disappearance of the intracranial vasosparm

SUMMARY:
The prevalence and clinical implications of prolonged cerebral vasospasm in patients with subarachnoid hemorrhage are unknown.

DETAILED DESCRIPTION:
The prevalence and clinical importance of prolonged cerebral vasospasm (after day 21 of bleeding) in patients with subarachnoid hemorrhage is unknown.

Objectives: To determine the prevalence and clinical relevance of prolonged vasospasm in patients with subarachnoid hemorrhage secondary to cerebral aneurysm.

A prospective and observational study was conducted. Adult patients with a diagnosis of subarcnoid hemorrhage CT scan or presence of blood in the cerebrospinal fluid were incorporated. Patients with vasospasm were followed daily with transcranial doppler. Those with technical impossibility to perform transcranial and pregnant Doppler were excluded. Day 0 was defined, the day of the last bleeding.

Evaluation: 1) It was considered in patients with prolonged vasospasm: whether or not it was associated with clinical manifestation (deterioration of the sensory or new neurological deficit) and 2) the magnitude of the vasospasm (mild, moderate or severe) was measured by transcranial doppler.

ELIGIBILITY:
Inclusion Criteria: Subarachnoid hemorrhage -

Exclusion Criteria: Pregnancy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid hemorrhage and vasospasm
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Clinical implication | 1 month
  Presence or not of neurological symptoms related to intracranial vasospasm (delayed cerebral ischemia)
Gravity of vasospasm by transcranial doppler | 1 month
  Mild, moderate and severe according to Aaslid scale

SECONDARY OUTCOMES:
Mortality assessment | six monts
  Mortality was assessed at hospital discharge and at six months

OTHER OUTCOMES:
Neurological recovery | six monts
  Neurological recovery at six months according to Glasgow outcome scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harders AG, Gilsbach JM. Time course of blood velocity changes related to vasospasm in the circle of Willis measured by transcranial Doppler ultrasound. J Neurosurg. 1987 May;66(5):718-28. doi: 10.3171/jns.1987.66.5.0718. PMID 3553456
- [Result] MASPES PE, MARINI G. Intracranial arterial spasm related to supraclinoid ruptured aneurysms. Acta Neurochir (Wien). 1962 Dec 12;10:630-8. doi: 10.1007/BF01406192. No abstract available. PMID 13933363
- [Result] Yamaguchi M, Bun T, Kuwahara T, Kitamura S. Very late-onset symptomatic cerebral vasospasm caused by a large residual aneurysmal subarachnoid hematoma--case report. Neurol Med Chir (Tokyo). 1999 Sep;39(9):677-80. doi: 10.2176/nmc.39.677. PMID 10563118
- [Result] Muller M, Schwerdtfeger K, Zieroth S. Assessment of middle cerebral artery diameter after aneurysmal subarachnoid hemorrhage by transcranial color-coded duplex sonography. Eur J Ultrasound. 2000 Mar;11(1):15-9. doi: 10.1016/s0929-8266(99)00066-x. PMID 10717509